CLINICAL TRIAL: NCT02673073
Title: Self-Awareness of Symptoms, Signs and Medical Compliance Using a Patient Diary in Heart Failure Management (AWARE-HF)
Brief Title: Self-Awareness of Symptoms, Signs and Medical Compliance Using a Patient Diary in Heart Failure Management
Acronym: AWARE-HF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, MD, PhD, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AWARE-HF
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Heart failure; patient's diary; self awareness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control_Education (Placebo Comparator): All patients will receive patient's information/education booklet on the heart failure including life style modification.
  Interventions: Other: Patient's education
- Intervention_Diary (Experimental): All patients will receive patient's information/education booklet on the heart failure including life style modification. In addition, patients also receive a patient's diary for self-recording of 6 parameters: body weight, blood pressure, heart rate, number of remaining pills, degree of pitting edema, and degree of dyspnea.
  Interventions: Other: Patient's diary

INTERVENTIONS:
Other: Patient's diary — Patients in the intervention arm will be educated to measure body weight, blood pressure, and heart rate every morning after using toilet. Number of remaining pills of the previous day is for the assessment of drug compliance. Degree of pitting edema is graded from 0 (no edema), 1 (mild), 2 (moderate), 3 (severe) and, degree of dyspnea is graded from 0, 1, 2, 3, corresponding to NYHA class I, II, III, and IV, respectively.
  Patients are instructed to visit or call the HF-outpatient clinic, when they have (i) body weight gain more than 1 kg/day or 2kg in 7 days;(ii) aggravation of pitting edema by one degree; (iii) aggravation of dyspnea by one grade.
  Arms: Intervention_Diary
Other: Patient's education — All patients will receive patient's information/education booklet on the heart failure including life style modification.
  Arms: Control_Education

SUMMARY:
Before a HF patient gets maximally decompensated and visit emergency department, most patients experience symptoms and signs of "on-going decompensation (or pre-decompensation)", which may not be noticed by the patients. If HF patients were aware of symptoms and signs of ADHF and received early intervention to stop the process of "on-going decompensation (or pre-decompensation)", it would be possible to reduce the rate of hospitalization for ADHF or death. Thus, self-awareness and self-examination of heart failure symptoms, signs and medical compliance using a patient diary in HF management may improve the outcomes in chronic stable HF patients. A patient diary with 6 parameters can serve this purpose: body weight, blood pressure, heart rate, drug compliance expressed as number of remaining pills of previous day, edema grade, and dyspnea grade.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older
* Patients admitted for acute heart failure and scheduled for discharge after medical stabilization
* Chronic stable heart failure patients with a history of hospitalization for AHF

Exclusion Criteria:

* Patients with limited cognitive function who cannot not perform self-recording (in case that the patient has a family member who can perform the recording, the patient can be rerolled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death or rehospitalization | 1 year
  Data on primary and secondary measures will be collected a trained study coordinator, using a standardized case report form.

SECONDARY OUTCOMES:
all-cause death | 1 year
cardiovascular death | 1 year
admission for acute heart failure | 1 year
drug compliance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jin Joo Park, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Retrum JH, Boggs J, Hersh A, Wright L, Main DS, Magid DJ, Allen LA. Patient-identified factors related to heart failure readmissions. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):171-7. doi: 10.1161/CIRCOUTCOMES.112.967356. Epub 2013 Feb 5. PMID 23386663
- [Background] Lee KS, Lennie TA, Warden S, Jacobs-Lawson JM, Moser DK. A comprehensive symptom diary intervention to improve outcomes in patients with HF: a pilot study. J Card Fail. 2013 Sep;19(9):647-54. doi: 10.1016/j.cardfail.2013.07.001. PMID 24054342
- [Background] Kato N, Kinugawa K, Nakayama E, Tsuji T, Kumagai Y, Imamura T, Maki H, Shiga T, Hatano M, Yao A, Miura C, Komuro I, Nagai R. Insufficient self-care is an independent risk factor for adverse clinical outcomes in Japanese patients with heart failure. Int Heart J. 2013;54(6):382-9. doi: 10.1536/ihj.54.382. PMID 24309448
- [Result] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Result] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602